CLINICAL TRIAL: NCT02051179
Title: Longitudinal Results of a 10-Year Clinical Trial of Repair of Amalgam Restorations
Acronym: REPAMLG
Status: Completed | Type: Observational
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Eduardo Fernandez, Prof. Eduardo Fernández Godoy, University of Chile
Other Study IDs: FOUCH 2012/10/2
Record Dates: First submitted 2014-01-25; First posted 2014-01-31 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2014-01

CONDITIONS: Unsatisfactory or Defective Restoration of Tooth
Keywords: Repair; Replacement; Dental Amalgam

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Replacement amalgam: Replacement The clinicians totally removed and replaced the defective restorations. After completing the cavity preparations, the tooth was restored with a new AM (Original D). Bonding agents and/or liners underneath the amalgam restorations were not used in this trial. Rubber dam isolation was used for all restorative treatments. .
- Repair Amalgam: The clinicians (PV and CM) used Carbide burs (330-010 Komet, Brasseler GmbH Co. Postfach 160.32631, Lemgo, Germany) to explore the defective margin, carious lesion or anatomic form of the restorations. Part of the restorative material adjacent to the defect was removed as an exploratory proceedure thus allowing a proper evaluation and subsequent diagnosis of the extent of the defect. Provided that the defect was limited and localized, the clinician then removed any defective tooth tissue. Mechanical retention was employed inside the existing AM restoration. Rubber dam isolation was used for this procedure. Repair of the restorations was carried out with a dispersed-phased amalgam (Original D, Wyckle Research Inc, Carson City, NV, USA).

SUMMARY:
The aim of this prospective, randomized clinical trial was to assess the effectiveness of repair of localized clinical defects of amalgam restorations that were initially scheduled for replacement of restorations. A cohort of 20 patients with 40 (Class I and Class II) amalgam restorations, that presented one or more clinical features that deviated from the ideal (Bravo or Charlie) according to USPHS criteria, were randomly assigned to either, the repair or replacement group: A: repair n= 19 and B: replacement n=21. Two examiners who had calibration exercised evaluated the restorations at baseline and ten years after according to seven parameters: marginal occlusal adaptation, anatomic form, surface roughness, marginal staining, contact, secondary caries, and luster

DETAILED DESCRIPTION:
Study Design A cohort of 20 patients between the ages of 18 to 80 years old (mean 26.5 years), female (58%) and male (42%), with 40 (Class I and Class II) amalgam restorations, that presented one or more clinical features that deviated from the ideal (Bravo or Charlie according to modified United States Public Health Service USPHS criteria). All of them were recruited at the Operative Dentistry Clinic at the Dental School, University of Chile. The protocol was approved by the Institutional Research Ethics Committee of the Dental School at the University of Chile (project PRI-ODO-0207), and all patients signed an informed consent form and completed a registration form.

Treatment Group Criteria: 40 defective restorations were evaluated in accordance with the modified USPHS criteria. Restorations with clinically diagnosed secondary caries (Charlie) or under-contoured or over-contoured anatomic form defects and restorations with marginal defects (Bravo) were randomly assigned (Random Number Generator, Microsoft Excel 97) to either, the repair or replacement group. Diagnosis of active secondary caries was done according to Ekstrand's criteria 31.

The groups were labeled A: repair n= 19 (Class I n=8 and Class II n=11) and B: replacement n=21 (Class I n=9 and Class II n=12).

Restorations Assessment and Outcome Measurements. The quality of the restorations was scored according to the modified USPHS criteria (Table 1) 32. Two examiners underwent calibration exercises (JM and EF, Cohen's Kappa inter-examiner coefficient 0.74 at baseline and 0.87 at ten years). The examiners assessed the restorations independently by direct visual and tactile examination (mouth mirror, number 5, Hu Friedy Mfg. Co. Inc., Chicago, IL, USA, and explorer, number 23, Hu Friedy) and indirectly by radiographic examination (Bite Wing) at baseline (immediately after treatment) and 10 years after treatment. The seven examined parameters were marginal occlusal adaptation (MA), anatomic form (A), surface roughness (R), Marginal staining (MS), occlusal contact (O), secondary caries (SC), and luster (L) (Table 1). If any difference was recorded between the two examiners, and if they did not reach an agreement, a third clinician, who also underwent calibration exercises (GM), made the final decision.

Treatment Group

A. Repair The clinicians (PV and CM) used Carbide burs (330-010 Komet, Brasseler GmbH Co. Postfach 160.32631, Lemgo, Germany) to explore the defective margin, carious lesion or anatomic form of the restorations. Part of the restorative material adjacent to the defect was removed as an exploratory proceedure thus allowing a proper evaluation and subsequent diagnosis of the extent of the defect. Provided that the defect was limited and localized, the clinician then removed any defective tooth tissue. Mechanical retention was employed inside the existing AM restoration. Rubber dam isolation was used for this procedure. Repair of the restorations was carried out with a dispersed-phased amalgam (Original D, Wyckle Research Inc, Carson City, NV, USA).

B. Replacement The clinicians totally removed and replaced the defective restorations. After completing the cavity preparations, the tooth was restored with a new AM (Original D). Bonding agents and/or liners underneath the amalgam restorations were not used in this trial. Rubber dam isolation was used for all restorative treatments. .

Patients were recalled after four and ten years after the restoration were placed for clinical assessment by the same examiners, applying the same criteria used at baseline. Failed restorations were removed from the study and treated according to their diagnosed needs.

Statistical analysis The ordinal dependent variable was changed in level of the modified USPHS criteria from the baseline value. The assigned score of each restoration reflected the worst result for any of the parameters. The results of each group in terms of degradation or upgrade were analyzed by Friedman range non-parametric test to compare the pre and postoperative conditions. Additionally, the performance of all groups was contrasted using the Mann Whitney test to determine the differences between the upgrade and downgrade of the restoration´s quality. The statistical significance was set at 95%, α=0.05 and β=0.80, SPSS15.0 (SPSS Inc, Chicago, IL) was used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* patients having at least one tooth with a localized marginal defective amalgam restoration(s) that was clinically determined to be suitable for repair, according to USPHS criteria
* patients with at least 20 teeth;
* restorations in functional occlusion with at least one opposing natural tooth;
* asymptomatic of post-operative sensitivity;
* with occlusal and proximal contact areas;
* patients older than 18 years; and
* patients who agreed and signed the informed consent form for participating in the study.

Exclusion Criteria:

* patients with contraindications for regular dental treatment based on their medical history
* patients who had special aesthetic needs that could not be solved by repair treatments
* patients with xerostomia and/or patients who were taking medication that significantly decreased salivary flow
* patients with high risk for caries
* patients with psychiatric or physical diseases, which interfered with oral hygiene

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A cohort of 20 patients between the ages of 18 to 80 years old (mean 26.5 years), female (58%) and male (42%), with 40 (Class I and Class II) amalgam restorations, that presented one or more clinical features that deviated from the ideal (Bravo or Charlie according to modified United States Public Health Service USPHS criteria). All of them were recruited at the Operative Dentistry Clinic at the Dental School, University of Chile
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2003-08; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Quality amalgam restorations | 10 years
  20 healthy voluteers with amalgam restorations , assesment of quality of amalgams by USPHS criterial

CONTACTS AND LOCATIONS:
Overall Officials: eduardo fernandez, Principal Investigator — University of Chile
Locations (1):
- Eduardo Fernández Godoy, Santiago, Chile

REFERENCES:
- [Result] Martin J, Fernandez E, Estay J, Gordan VV, Mjor IA, Moncada G. Management of Class I and Class II Amalgam Restorations with Localized Defects: Five-Year Results. Int J Dent. 2013;2013:450260. doi: 10.1155/2013/450260. Epub 2013 Jan 28. PMID 23431302
- [Result] Martin J, Fernandez E, Estay J, Gordan VV, Mjor IA, Moncada G. Minimal invasive treatment for defective restorations: five-year results using sealants. Oper Dent. 2013 Mar-Apr;38(2):125-33. doi: 10.2341/12-062C. Epub 2012 Jul 11. PMID 22788726
- [Result] Fernandez EM, Martin JA, Angel PA, Mjor IA, Gordan VV, Moncada GA. Survival rate of sealed, refurbished and repaired defective restorations: 4-year follow-up. Braz Dent J. 2011;22(2):134-9. doi: 10.1590/s0103-64402011000200008. PMID 21537587
- [Result] Moncada G, Martin J, Fernandez E, Hempel MC, Mjor IA, Gordan VV. Sealing, refurbishment and repair of Class I and Class II defective restorations: a three-year clinical trial. J Am Dent Assoc. 2009 Apr;140(4):425-32. doi: 10.14219/jada.archive.2009.0191. PMID 19339531
- [Result] Moncada G, Fernandez E, Martin J, Arancibia C, Mjor IA, Gordan VV. Increasing the longevity of restorations by minimal intervention: a two-year clinical trial. Oper Dent. 2008 May-Jun;33(3):258-64. doi: 10.2341/07-113. PMID 18505215
- [Result] Moncada GC, Martin J, Fernandez E, Vildosola PG, Caamano C, Caro MJ, Mjor IA, Gordan VV. Alternative treatments for resin-based composite and amalgam restorations with marginal defects: a 12-month clinical trial. Gen Dent. 2006 Sep-Oct;54(5):314-8. PMID 17004564